CLINICAL TRIAL: NCT04960007
Title: Comparison of the Swallowing Functions of the Sarcopenia and Dynapenia Patients
Brief Title: Comparison of the Swallowing Functions in Sarcopenia and Dynapenia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Sevgi Atar, Specialist, MD, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 261
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Sarcopenia; Dysphagia; Swallowing Disorder
Keywords: sarcopenia; dynapenia; swallowing; deglutition; dysphagia
MeSH Terms: conditions — Sarcopenia; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Sarcopenia patients.
- Group B: Dynapenia patients.
- Group C: Age and gender matched non-sarcopenia and non-dynapenia patients.

SUMMARY:
The purpose of the study to investigate the comparison of the swallowing functions of the sarcopenia and dynapenia in older patients

DETAILED DESCRIPTION:
Sarcopenia is a geriatric syndrome; from skeletal muscle, and in its usefulness. Dynapenia is a picture of sarcopenia without measurable muscle mass. It has been shown that dysphagia complaints are more common in patients with sarcopenia than in the normal population, but a comparison with patients with dynapenia has not been made to the best of our knowledge. According to the algorithm of The International Society of Physical and Rehabilitation Medicine (ISPRM), experts in the special interest group on sarcopenia, in the routine examination of patients aged 60-90 years who applied to the Physical Medicine and Rehabilitation outpatient clinic with complaints of decreased muscle function, weakness, and slow movement, or "sarcopenia" or Patients with "dynapenia" and patients without Sarcopenia disease who volunteered to participate in the study will be included in the order of application to the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60-90 years
* Sarcopenia and dynapenia patients in study groups
* Non- sarcopenia and non-dynapenia patients in control groups
* Patients who were accept to consent form

Exclusion Criteria:

* Severe sarcopenia patients
* Cognitive limitations
* Out of age 60-90 years old
* Patients who were not accept to consent form

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were 60-90 years old.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2021-08-27 (Estimated); Study Completion 2021-08-27 (Estimated)

PRIMARY OUTCOMES:
The values of Pharyngeal Residue Severity | Baseline
  It was assessed with Fiberoptic Endoscopic Evaluation of Swallowing. Fiberoptic Endoscopic Evaluation of Swallowing results were scored on Yale Pharyngeal Residue Severity Rating scale. The scores of scale were none, trace, mild, moderate, and severe. The high-grade symptom scores were worst, low scores were good swallowing functions.
The values of penetration and aspiration | Baseline
  It was assessed with Fiberoptic Endoscopic Evaluation of Swallowing. Fiberoptic Endoscopic Evaluation of Swallowing results were scored on the Penetration and aspiration scale. The scores of scale were between 1-8 points. The high points were worst, low points were good swallowing functions.
The evaluation of eating and swallowing functions | Baseline
  They were assessed by Eating Assessment Tool in participants. Composite Score ranges from 0 ( good) to 4 (worst). The minimum total score was 0 and the maximum total score was 40. The cut-off value was 3 points. High scores show worst eating and swallowing functions, and low quality of life.
The evaluation of depression | Baseline
  They were assessed by Geriatric Depression Scale in participants. The scores between 0-10 were no depression, between 11-13 points were probably depression, and higher of 14 points were exact depression.
The values of muscle strength | Baseline
  They were assessed as newton by hand grip device.
The values of muscle mass | Baseline
  The diameters of tigh were measured with tailor meter by a Physical Medicine and Rehabilitation professionals (measure unit is cm).

SECONDARY OUTCOMES:
Mean of demographic | Baseline
  Age, gender, history of smoke, history of morbidities, diagnosis, stage, were noted

CONTACTS AND LOCATIONS:
Overall Officials: yavuz atar, Asso Prof,MD, Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Prof Dr Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Firat Ozer F, Akin S, Soysal T, Gokcekuyu BM, Erturk Zararsiz G. Relationship Between Dysphagia and Sarcopenia with Comprehensive Geriatric Evaluation. Dysphagia. 2021 Feb;36(1):140-146. doi: 10.1007/s00455-020-10120-3. Epub 2020 Apr 27. PMID 32342177
- [Background] Kara M, Kaymak B, Frontera W, Ata AM, Ricci V, Ekiz T, Chang KV, Han DS, Michail X, Quittan M, Lim JY, Bean JF, Franchignoni F, Ozcakar L. Diagnosing sarcopenia: Functional perspectives and a new algorithm from the ISarcoPRM. J Rehabil Med. 2021 Jun 21;53(6):jrm00209. doi: 10.2340/16501977-2851. PMID 34121127
- [Background] Chen YC, Chen PY, Wang YC, Wang TG, Han DS. Decreased swallowing function in the sarcopenic elderly without clinical dysphagia: a cross-sectional study. BMC Geriatr. 2020 Oct 21;20(1):419. doi: 10.1186/s12877-020-01832-0. PMID 33087067